CLINICAL TRIAL: NCT04914208
Title: Effect of Wearing Face Masks on Oral Health
Brief Title: Effect of Wearing Face Masks on Salivary Parameters and Halitosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Göttingen (Other)
Responsible Party: Principal Investigator, Philipp Kanzow, PD Dr. med. dent., Dr. rer. medic., Senior Dental Practitioner, University Medical Center Goettingen
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: FaceMasks-Halitosis; 30/2/21 (Other: Local Ethics Commission); 2021-01521 (Other: UMG study center)
Record Dates: First submitted 2021-05-30; First posted 2021-06-04 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-02

CONDITIONS: Dry Mouth; Halitosis
MeSH Terms: conditions — Xerostomia; Halitosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Wearing a face mask for 4 hours (Active Comparator): Participants are wearing different kinds of face masks for 4 hours each. Masks are worn on different days and the order is randomly assigned.
  Interventions: Device: DIY face mask; Device: Surgical face mask; Device: FFP2 respirator mask; Other: Use of fluoridated toothpaste
- 4 hours without wearing a face mask (Other): Participants do not wear any face mask for 4 hours.
  Interventions: Other: Waiting for 4 hours without wearing a mask; Other: Use of fluoridated toothpaste

INTERVENTIONS:
Device: DIY face mask — Participants are wearing a DIY face mask for 4 hours (beginning between 8 and 9 a.m.). The correct fit of the face mask is checked by the study officials and corrected if necessary.
  Arms: Wearing a face mask for 4 hours
Device: Surgical face mask — Participants are wearing a surgical face mask for 4 hours (beginning between 8 and 9 a.m.). The correct fit of the face mask is checked by the study officials and corrected if necessary.
  Arms: Wearing a face mask for 4 hours
Device: FFP2 respirator mask — Participants are wearing a FFP2 respirator mask for 4 hours (beginning between 8 and 9 a.m.). The correct fit of the face mask is checked by the study officials and corrected if necessary.
  Arms: Wearing a face mask for 4 hours
Other: Waiting for 4 hours without wearing a mask — Participants do not wear any face mask for 4 hours (beginning between 8 and 9 a.m.).
  Arms: 4 hours without wearing a face mask
Other: Use of fluoridated toothpaste — Participants use fluoridated toothpaste.

SUMMARY:
During the current COVID-19 pandemic, the use of face masks is recommended / mandatory to prevent infection. Patients and students have reported to experience limitations in their oral health-related quality of life, especially with regard to the occurrence of dry mouth and halitosis, while wearing face masks.

Scientific studies regarding the effects of face masks have so far focused exclusively on medical staff. Studies among the general population are not yet available, but are of interest as dry mouth is a risk factor for dental diseases (e.g., caries, erosion).

Therefore, the present study aims at measuring the effect of wearing different face masks on salivary parameters (unstimulated and stimulated saliva flow rate, pH, buffer capacity) and halitosis (volatile sulphur compounds).

ELIGIBILITY:
Inclusion Criteria:

* Oral healthy adult volunteers who are able to give written consent

Exclusion Criteria:

* Non-fulfillment of the inclusion criteria
* Denied access to the University Medical Center Goettingen at the Corona screening
* Exemption from wearing a face mask for medical reasons
* Medical reasons hindering participants from refraining eating and drinking prior (except for water) or during the visits
* Hyposalivation / xerostomia (unstimulated saliva < 0.3 mL/min, stimulated saliva < 0.7 mL/min)
* Refusal to use fluoridated toothpastes
* Smoking

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-09-28 (Actual); Primary Completion 2022-04-08 (Actual); Study Completion 2022-04-08 (Actual)

PRIMARY OUTCOMES:
Determination of unstimulated saliva flow rate | Each day, prior (between 8 and 9 a.m.) and after wearing a face mask for 4 hours or 4 hours without wearing any mask. Saliva samples are collected for 5 min each.
  mL/min

SECONDARY OUTCOMES:
Determination of stimulated saliva flow rate | Each day, prior (between 8 and 9 a.m.) and after wearing a face mask for 4 hours or 4 hours without wearing any mask. Stimulated saliva samples are collected for 5 min while chewing a paraffin pellet.
  mL/min
Determination of unstimulated and stimulated saliva pH | Each day, prior (between 8 and 9 a.m.) and after wearing a face mask for 4 hours or 4 hours without wearing any mask. Saliva samples are collected for 5 min each. Stimulated saliva samples are collected while chewing a paraffin pellet.
  pH
Determination of unstimulated and stimulated salivary buffer capacity | Each day, prior (between 8 and 9 a.m.) and after wearing a face mask for 4 hours or 4 hours without wearing any mask. Saliva samples are collected for 5 min each. Stimulated saliva samples are collected while chewing a paraffin pellet.
  pH
Determination of volatile sulphur compounds (VSC) | Each day, prior (between 8 and 9 a.m.) and after wearing a face mask for 4 hours or 4 hours without wearing any mask.
  ppm

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center Goettingen, Dept. of Preventive Dentistry, Periodontology and Cariology, Göttingen, Lower Saxony, Germany

REFERENCES:
- [Background] Farronato M, Boccalari E, Del Rosso E, Lanteri V, Mulder R, Maspero C. A Scoping Review of Respirator Literature and a Survey among Dental Professionals. Int J Environ Res Public Health. 2020 Aug 17;17(16):5968. doi: 10.3390/ijerph17165968. PMID 32824564
- [Background] Rebmann T, Carrico R, Wang J. Physiologic and other effects and compliance with long-term respirator use among medical intensive care unit nurses. Am J Infect Control. 2013 Dec;41(12):1218-23. doi: 10.1016/j.ajic.2013.02.017. Epub 2013 Jun 12. PMID 23768438
- [Background] Shenal BV, Radonovich LJ Jr, Cheng J, Hodgson M, Bender BS. Discomfort and exertion associated with prolonged wear of respiratory protection in a health care setting. J Occup Environ Hyg. 2012;9(1):59-64. doi: 10.1080/15459624.2012.635133. PMID 22168256
- [Result] Kanzow P, Rammert LS, Rohland B, Barke S, Placzek M, Wiegand A. Effect of face masks on salivary parameters and halitosis: Randomized controlled crossover trial. J Oral Pathol Med. 2023 Jan;52(1):56-62. doi: 10.1111/jop.13390. Epub 2022 Dec 13. PMID 36459058